CLINICAL TRIAL: NCT00144378
Title: Randomized Phase III Study With Irinotecan+Best Supportive Care Versus Only Best Supportive Care as Second Line Therapy for Metastatic Gastric Cancer
Brief Title: Irinotecan Versus Only Best Supportive Care for Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: irinotecan vs. bsc
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Stomach Neoplasm; Neoplasm Metastasis
Keywords: gastric cancer; metastatic; irinotecan
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Irinotecan

INTERVENTIONS:
Drug: Irinotecan

SUMMARY:
The median survival at progression after first-line chemotherapy for metastatic gastric cancer is about 2.5 months. There are no data which a possible benefit of second line therapy. for this reason a trial which investigates a possible benefit or chemotherapy compared to best supportive care as second line treatment is urgently necessary.

Irinotecan shows response rates of 20% in the first line therapy with high rates od disease stabilization. There are few trials investigating irinotecan in the second line setting. Response rates of 20% are reported in tis setting. Irinotecan is supplied without costs from the company Pfizer.

DETAILED DESCRIPTION:
Metastatic gastric cancer, progressive disease after one palliative chemotherapy

Arm A:

Irinotecan 250/350 mg/m2 q3w

1. Cycle:250mg/m2/ 30min
2. Cycle:If no toxicity>2° CTC, nor Leuko-thrombopenia>3° occured, dose is increased to 350mg/m2 Arm B. Best supportive care

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven adenocarcinoma of stomach or the gastro-esophageal junction
* Patient with distant metastases laparoscopically proven operative incurability of an locally advanced gastric cancer or patient with a tumor recurrence after gastrectomy
* Patient with progressive disease under a palliative first-line chemotherapy or progressive disease within 6 months after termination of a first-line chemotherapy, defined as objective progression by imaging techniques according to WHO criteria
* Age 18 and 75 years
* Sufficient liver function, defined as serum-bilirubin <1,5 mg/dl (1,5 upper normal limit), ALT und AST < 3x upper normal limit
* Sufficient renal function, defined as serum creatinine < 1,25 x upper normal limit or creatinine clearance >60ml/min calculated according to Crockroft-Gault
* Contraction for patient with reproductive potential
* Karnofsky-Index >60%
* Measurable or evaluable tumor manifestation

Exclusion Criteria:

* Tumor progression later than 6 months after termination of first-line chemotherapy
* KI 50% or less
* Patient who have already received a second line chemotherapy for the metastatic setting (adjuvant chemotherapy and one line of palliative chemotherapy os allowed, biologic prior therapies are allowed)
* Prior or current second malignancy despite of basal carcinoma of the skin and curatively treated carcinoma in situ of the cervix
* Uncontrolled infection
* CNS metastases
* Other severe medical illness
* Prior major surgery less than 2 weeks ago
* Parallel treatment with another experimental therapy
* Parallel treatment with another therapy aiming at tumor reduction
* Chronic diarrhea, subileus
* Chronic inflammatory bowel disease or intestinal obstruction
* Pretreatment with irinotecan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2002-10

PRIMARY OUTCOMES:
median survival

SECONDARY OUTCOMES:
quality of life, response rates, time to tumor progression, toxicity

CONTACTS AND LOCATIONS:
Overall Officials: P Reichardt MD PhD, Principal Investigator — Charité, University,Campus Virchow Klinikum, Dep. of Hematology and Oncology,Berlin; PC Thuss-Patience MD PhD, Principal Investigator — Charité, University,Campus Virchow Klinikum,Dep. of Hematology and Oncology
Locations (1):
- Charité,Universitätsmedizin Berlin, Campus Virchow Klinikum, Dep. orf Hematology and Oncology,, Berlin, Germany

REFERENCES:
- [Derived] Thuss-Patience PC, Kretzschmar A, Bichev D, Deist T, Hinke A, Breithaupt K, Dogan Y, Gebauer B, Schumacher G, Reichardt P. Survival advantage for irinotecan versus best supportive care as second-line chemotherapy in gastric cancer--a randomised phase III study of the Arbeitsgemeinschaft Internistische Onkologie (AIO). Eur J Cancer. 2011 Oct;47(15):2306-14. doi: 10.1016/j.ejca.2011.06.002. PMID 21742485